CLINICAL TRIAL: NCT07200089
Title: A Double-blind, Placebo-controlled Phase Ib Study Evaluating the Safety and Toxicity of Recombinant Human IL-7 (NT-I7) in Relapsed/Refractory Multiple Myeloma Following BCMA CAR-T Therapy (Cilta-cel)
Brief Title: Recombinant Human IL-7 (NT-I7) in Relapsed/Refractory Multiple Myeloma Following BCMA CAR-T Therapy (Cilta-cel)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: NeoImmuneTech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25-x122
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
Keywords: Cytokines; Interleukin-7; Cellular therapy; Chimeric antigen receptor T cell therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — efineptakin alfa; B-Cell Maturation Antigen; bis(3-bis(4-chlorophenyl)methyl-4-dimethylaminophenyl)amine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: NT-I7 (Experimental): Patients randomized to the intervention arm will receive 720 μg/kg NT-I7 intramuscularly on Day 14 and a second dose on Day 35 after BCMA CAR-T infusion.
- Control: Placebo (Active Comparator): Patients randomized to the control arm will receive a placebo on Days 14 and 35.
  Interventions: Drug: Placebo; Biological: B-cell Maturation Antigen (BCMA) CART-T therapy

INTERVENTIONS:
Drug: NT-I7 — NT-I7 will be supplied by NeoImmuneTech Inc
  Other Names: Recombinant human IL-7
Drug: Placebo — Placebo will be supplied by NeoImmuneTech Inc
  Arms: Control: Placebo
Biological: B-cell Maturation Antigen (BCMA) CART-T therapy — Standard of care
  Arms: Control: Placebo

SUMMARY:
CAR-T cell therapy is an emerging treatment modality in relapsed and refractory multiple myeloma (MM). CAR-T therapy in MM relies on directing autologous T-cells to detect and clear myeloma cells expressing B-cell Maturation Antigen (BCMA). While BCMA CAR-T cell-treated patients achieve an excellent overall response rate, their response is often not durable. NT-I7 promotes CAR-T cell expansion and efficacy in pre-clinical lymphoma models. In patients receiving CD19-directed CAR-T therapy for lymphoma, NT-I7 augmented CAR-T expansion while being safe and tolerable. The impact of NT-I7 on BCMA CAR-T cells in multiple myeloma is unknown.

This is a two-arm, double blind, placebo-controlled, randomized, single-site phase Ib study testing the safety and toxicity of adding NT-I7 to BCMA CAR-T therapy in patients with relapsed and refractory multiple myeloma. The hypothesis is that NT-I7 will promote CAR-T expansion and persistence which will enhance clearance of MM, while maintaining a favorable safety and toxicity profile. Patients receiving standard of care BCMA CAR-T (Cilta-cel) will be randomized to either NT-I7 or placebo. Correlative studies will evaluate CAR-T cell expansion, persistence, immune-phenotype, function and correlate with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma with measurable disease by IMWG criteria.
* Eligible for standard of care BCMA CAR-T cell therapy.
* Life expectancy ≥ 12 weeks per assessment from the enrolling physician.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Adequate organ function as defined below:

  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine clearance > 30 mL/min by Cockcroft-Gault
* The effects of NT-I7 on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception prior to study entry until 90 days after completion of NT-I7 therapy/placebo (corresponding to Day 125 post CAR-T). Should a woman become pregnant or suspect she is pregnant while participating in this study or should a man suspect he has fathered a child, s/he must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Received prior BCMA-directed therapy.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial.
* Currently receiving or have received any other investigational agents within 14 days prior to CAR-T infusion.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to NT-I7or other agents used in the study.
* Uncontrolled intercurrent illness including but not limited to: ongoing or active infection (bacterial, fungal, viral, or tuberculosis, including known hepatitis A, B, or C, or HIV (testing not required)), symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia (except well-controlled atrial fibrillation). Patients with a known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Function Classification; to be eligible for this trial, patients should be a class 2B or better.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to starting CAR-T therapy.
* Receipt of live, attenuated vaccine within 30 days prior to first day of treatment.
* Had an allogeneic tissue/solid organ transplant or allogeneic stem cell transplant.
* Not able to receive subcutaneous therapy.
* Prior history of T cell malignancy.
* Prior history of congenital immunodeficiency syndrome.
* Prior history of autoimmune disease with significant disease activity in the past 2 years, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, Sézary syndrome, vasculitis or glomerulonephritis, Bell's palsy, Guillain-Barré syndrome, or multiple sclerosis.
* Prior history of plasma cell leukemia, systemic amyloidosis, POEMS syndrome, or multiple myeloma with CNS involvement.
* Planning to start maintenance therapy prior to Day 100 post-CAR-T therapy.
* A history of clinically significant pulmonary disorders, such as severe asthma, severe COPD, restrictive lung disease, symptomatic pulmonary embolism within 3 months prior to study enrollment, or active or prior interstitial lung disease/pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-10-10 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of non-hematologic grade ≥3 treatment-related AEs (excluding expected conditioning-related AEs) | From Day 14 to Day 100
  Graded per CTCAE v 5.0.

SECONDARY OUTCOMES:
MRD negativity by clonoSEQ (10^5 cutoff) | At Day 100
MRD negativity by clonoSEQ (10^6 cutoff) | At Day 100
Number of participants with stringent complete response (sCR) by IMWG criteria | At Day 100
  * Stringent complete response requires all of the following:
    * CR as defined below
    * Normal free light chain ratio (0.26-1.65)
    * Absence of clonal cells in the bone marrow by immunohistochemistry or immunofluorescence
  * Complete response (CR) requires all of the following:
    * Negative immunofixation on the serum and urine
    * <5% plasma cells in the bone marrow aspirate
    * Disappearance of any soft tissue plasmacytomas
    * Normalization of the serum free light chain ratio in patients who lack measurable M protein in the serum and urine at baseline
Progression-free survival (PFS) | At Day 365
  * PFS is defined as the length of time between randomization and disease progression or death from any cause.
  * Progressive disease per IMWG criteria.
Number of participants with Grade ≥2 CRS and ICANS according to ASTCT consensus grading | From Day 0 through Day 100
Number of participants with Grade ≥3 CRS and ICANS according to ASTCT consensus grading | From Day 0 through Day 100
Rate of non-relapse mortality (NRM) | By Day 365
  For the purposes of this study, NRM is death following CAR-T cell infusion without evidence of progressive myeloma.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Slade, M.D., M.S.C.I, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient level data may be shared following publication of the manuscript analyzing the primary endpoint of this study.
Supporting Information: Study Protocol, SAP
Time Frame: Up to 5 years following trial completion.
Access Criteria: Interested researchers seeking access to de-identified data related to this trial should contact the principal investigator at sladem@wustl.edu. Requests will be considered on a case-by-case basis.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu